CLINICAL TRIAL: NCT05220449
Title: Individualized Brain Stimulation to Improve Functional Rehabilitation in Two Models of Sensorimotor Disorders: Stroke and Parkinson's Disease
Brief Title: Re-Orchestration of Interregional Oscillatory Activity to Promote Visual Recovery
Acronym: R4V
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ecole Polytechnique Fédérale de Lausanne (Other)
Responsible Party: Principal Investigator, Estelle Raffin, Teaching and Research Associate, Ecole Polytechnique Fédérale de Lausanne
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-01761
Record Dates: First submitted 2021-11-30; First posted 2022-02-02 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Visual Impairment; Stroke; Parkinson Disease
Keywords: Stroke; Visual field; Oscillations; tACS; Parkinson's Disease
MeSH Terms: conditions — Vision Disorders; Stroke; Parkinson Disease

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Double (Participant & Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cf-tACS (V1-Alpha_V5-Gamma) (Active Comparator)
  Interventions: Other: Cross-frequency dual-site tACS
- Cf-tACS (V1-Gamma_V5-Alpha) (Experimental)
  Interventions: Other: Cross-frequency dual-site tACS

INTERVENTIONS:
Other: Cross-frequency dual-site tACS — Dual site transcranial alternating current stimulation over the primary visual cortex (V1) and the mediotemporal cortex (MT/V5) using two different stimulation frequencies (Alpha and Gamma)

SUMMARY:
This project assesses the effect of bifocal cross-frequency transcranial alternating current stimulation (tACS) combined with visual training to improve visual recovery and orchestrated oscillatory activity in stroke patients suffering from visual field defects.

ELIGIBILITY:
Inclusion Criteria:

1. the patient can consent for themselves;
2. age 18+ years old;
3. at least 7 days since diagnosis "stroke".
4. Patients should demonstrate a clear deficit in either simple or complex visual perception in portions of their visual field

Exclusion Criteria:

1. Diminished capacity to consent;
2. Pregnancy
3. Known or suspected non-compliance, drug or alcohol abuse
4. Inability to follow the procedures of the study, e.g., due to language problems, psychological disorders, dementia, etc. of the participant,
5. Non-compliance to the instructions of the experimenter or an inappropriate behavior hindering the normal progress of the experiment.
6. Previous enrolment into the current study
7. Exclusion criteria of MRI, tACS, TMS
8. Use of psychoactive medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Changes in visual field functions | Measured at baseline (i.e. before the first day of intervention), and post intervention (i.e., after the last day of intervention)
  Comparison of the systematic measurement of the visual field using Humphrey perimetry

SECONDARY OUTCOMES:
Changes in motion discrimination and integration performances | Measured at baseline (i.e. before the first day of intervention), and post intervention (i.e., after the last day of intervention)
  Comparison of the motion coherence threshold extracted from a two forced-choice direction discrimination task
Changes in inter-areal cross-frequency interaction | Measured at baseline (i.e. before the first day of intervention), and post intervention (i.e., after the last day of intervention)
  Comparison of the inter-areal Alpha-Gamma coupling using electroencephalography recordings
Changes in visual tracts integrity | Measured at baseline (i.e. before the first day of intervention), and post intervention (i.e., after the last day of intervention)
  Comparison of the diffusion weigted imaging-based tractography of the main visual tracts
Changes in functional connectivity within the broad visual network | Measured at baseline (i.e. before the first day of intervention), and post intervention (i.e., after the last day of intervention)
  Functional MRI based connectivity analyses using DCM or graph theory will perfomed

CONTACTS AND LOCATIONS:
Locations (1):
- Campus Biotech, EPFL, Geneva, Switzerland